CLINICAL TRIAL: NCT03826693
Title: Efficacy of Nitrous Oxide in OCD: Pilot Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Peter J van Roessel, MD PhD, Clinical Associate Professor, Department of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48077
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; nitrous oxide
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Nitrous Oxide; Nitrogen

STUDY DESIGN:
Intervention Model Description: placebo-controlled 2:1 randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Nitrous Oxide (Experimental): OCD participants in this arm will receive 50%oxygen/50% nitrous oxide admixture for 60 minutes.
  Interventions: Drug: Nitrous Oxide
- Control: Nitrogen (Placebo Comparator): OCD participants in this arm will receive 50%oxygen/50% nitrogen admixture for 60 minutes.
  Interventions: Drug: Nitrogen

INTERVENTIONS:
Drug: Nitrous Oxide — OCD participants in this arm will receive 50%oxygen/50% nitrous oxide admixture for 60 minutes.
  Arms: Experimental: Nitrous Oxide
Drug: Nitrogen — OCD participants in this arm will receive 50%oxygen/50% nitrogen admixture for 60 minutes.
  Arms: Control: Nitrogen

SUMMARY:
This study investigates whether the commonly used and well-tolerated inhaled anesthetic nitrous oxide can rapidly improve symptoms of OCD.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a chronic and disabling disorder characterized by recurrent intrusive thoughts and associated compulsive behaviors that is estimated to affect more than 3 million individuals in the US each year.

This study seeks to explore whether a single inhalation of nitrous oxide gas may bring about rapid symptom relief in OCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Primary diagnosis of OCD
* Sufficient severity of OCD symptoms
* Ability to tolerate a treatment-free period
* Capacity to provide informed consent

Exclusion Criteria:

* Psychiatric or medical conditions that make participation unsafe
* Pregnant or nursing females
* Concurrent use of any medications that might increase the risk of participation (e.g. drug interactions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-04-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in the severity of OCD symptoms as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | 1 week
  Improvement in OCD severity is measured by the YBOCS (Yale Brown Obsessive-Compulsive Scale), a gold standard measure of obsessions and compulsions. For the YBOCS the minimum units are 0 and Maximum units on the total scale are 40. The higher the number on the YBOCS, the more severe the symptoms. Response is defined as at least a 35% reduction on the YBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J van Roessel, MD, PhD, Principal Investigator — Stanford Univeristy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford Medicine Faculty Page — https://med.stanford.edu/profiles/peter-van-roessel
- See also: Rodriguez Lab Website — https://rodriguezlab.stanford.edu